# CLINICAL EVALUATION OF THREE DIFFERENT BIOACTIVE RESTORATIVE MATERIALS IN CERVICAL CARIOUS LESIONS IN HIGH CARIES RISK PATIENTS: A Randomized Controlled Clinical Trial

#### Protocol submitted to

Faculty of Dentistry, Cairo University for partial fulfillment of the requirements **for the PhD Degree** in Restorative and Esthetic Dentistry.

## By

#### Ahmed Abdul Monsif Abdul Mohsen Abdul Aziz

ID: 14422022532609
Theme .Objective code: CONS 3.7.5
BDS 2011, Faculty of Dentistry, MUST University
MSc. 2019, Faculty of Dentistry, Al-Azhar University
2024

Code: CONS 3.7.5

Supervisors' signature signature

Head of department's

- 1- Ashraf nasr
- 2- Dr. Yehia Hafez

Date



# Medical Biostatistics Unit review report for sample size calculation



#### **Individual Details**

First Name: Ahmed

Surname: Abdul monsif

Email address: ahmed.monsif@dentistry.cu.edu.eg

## **Department \***

**Conservative dentistry department** 

## Main Supervisor Details (if applicable)

Prof. Dr. Ashraf Nasr

Email address: ashraf.nasr@dentistry.cu.edu.eg

#### **Research Information**

Research title: CLINICAL EVALUATION OF THREE DIFFERENT BIOACTIVE RESTORATIVE MATERIALS IN CERVICAL CARIOUS LESIONS IN HIGH CARIES

RISK PATIENTS: A Randomized Controlled Clinical Trial

**Research question**: Will the three different bioactive restorative materials have the same clinical performance in cervical carious lesions in high caries risk patients over eighteen months of follow-up?

## Complete items used in sample size calculated \*

- The outcome used: Post operative hyper sensitivity (after 12 months)
- Values used for outcome: Proportions
- Entry 1: (estimated) 0.675 for I1 and I2
- Entry 2: 0.975
- Alpha level of significance: 0.05 (5%)
- Effect size: minimal clinically important difference of 30%
- Power of the study: 80%
- Statistical test used: Z test for two independent proportions
- The calculated sample size: 24 per group
- Increased number for anticipated missing data (10%): 27 per group

\* Date of submission: / / 2024 Date of approval: / /2024

Vice Dean for Postgraduate affairs and research